CLINICAL TRIAL: NCT07268144
Title: Effectiveness of a Supervised University-Based Physical Activity and Health Education Program on Lifestyle and Psychological Well-being: A Controlled Educational Intervention Study
Brief Title: Effectiveness of a Supervised University-Based Physical Activity and Health Education Program on Lifestyle and Psychological Well-being (Ponte en Forma)
Acronym: PONTE-FORMA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundacin Biomedica Galicia Sur (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PonteEnForma-UVIGO-2016; 2016/567 (Other: Ethics Committee Approval)
Record Dates: First submitted 2025-11-20; First posted 2025-12-05 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-12

CONDITIONS: Healthy Lifestyle; Cardiovascular Risk Factors; Sedentary Behavior; Psychological Well-being; Health Promotion
Keywords: University health promotion; Physical activity intervention; Mediterranean diet adherence; Lifestyle behavior change; Psychological well-being; Self-esteem; Emotional intelligence; Non-communicable diseases prevention; Young adults; Controlled educational intervention
MeSH Terms: conditions — Sedentary Behavior; Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: This study used a parallel-group, controlled educational intervention design. Participants were assigned to either the "Ponte en Forma" supervised physical activity and lifestyle counseling program (intervention group) or to a control group performing unsupervised exercise at the university facilities. Allocation was non-randomized and based on voluntary program enrollment.
Masking Description: Not applicable. Due to the nature of the educational and physical activity intervention, neither participants nor study staff could be blinded to group assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Arm - Ponte en Forma Program (Experimental): Participants in this group took part in the "Ponte en Forma" supervised physical activity and health education program conducted at the University of Vigo (Campus of Ourense). The program lasted four months and combined supervised exercise sessions three times per week with biweekly group or individual counseling on nutrition, tobacco and alcohol prevention, and emotional well-being. Attendance of at least 75% of sessions was considered adherent.
  Interventions: Behavioral: Ponte en Forma Program
- Control Arm - Usual Unsupervised Activity (No Intervention): Participants in the control group continued their usual unsupervised physical activity at the university sports facilities. They received only a written leaflet summarizing general recommendations on healthy diet, regular exercise, and avoidance of tobacco and alcohol, with no individualized supervision or follow-up.

INTERVENTIONS:
Behavioral: Ponte en Forma Program — A structured behavioral intervention combining supervised physical training and lifestyle education over a four-month period. The intervention included:
  Supervised exercise three times per week, integrating aerobic, strength, flexibility, and balance components adapted to individual fitness levels.
  Biweekly counseling sessions on healthy eating, adherence to the Mediterranean diet, prevention of tobacco and alcohol use, and emotional well-being strategies.
  Conducted by qualified sports science professionals and health educators. Other Name(s): University-based health promotion program
  Arms: Intervention Arm - Ponte en Forma Program

SUMMARY:
This study evaluates the effectiveness of a structured, supervised university-based program that combines physical activity and health education to promote healthy lifestyle behaviors and psychological well-being. The program, called Ponte en Forma, is implemented at the University of Vigo (Campus of Ourense, Spain) as part of its institutional health promotion strategy.

Adult participants (students, university staff, and community members) are allocated either to an intervention group, which takes part in the supervised Ponte en Forma program, or to a control group, which continues their usual unsupervised exercise routine. The intervention lasts four months and includes three weekly supervised exercise sessions plus biweekly counseling focused on healthy eating, prevention of tobacco and alcohol use, and emotional well-being.

The main outcomes assessed include body mass index (BMI), blood pressure, resting heart rate, and adherence to the Mediterranean diet. Secondary outcomes include self-esteem, emotional intelligence, health-related quality of life, and lifestyle habits.

DETAILED DESCRIPTION:
The Ponte en Forma program is a university-based health promotion initiative designed to improve physical, dietary, and psychological health through a combination of supervised exercise and lifestyle counseling. The program is implemented at the University of Vigo (Campus of Ourense, Spain) during the 2016-2017 academic year.

Study Design

This is a quasi-experimental, non-randomized, controlled intervention study. Participants are users of the University Sports Service. The intervention group participates in the supervised Ponte en Forma program, while the control group continues their regular unsupervised exercise activities. Allocation is based on type of enrollment and participant preference.

Intervention Details

The program includes three weekly sessions of supervised physical activity (aerobic, strength, flexibility, and balance training) and biweekly group or individual counseling sessions. Counseling addresses nutrition and the Mediterranean diet, avoidance of tobacco and alcohol consumption, and strategies for emotional well-being.

Outcome Measures

Primary outcomes:

Body Mass Index (BMI)

Systolic and diastolic blood pressure

Resting heart rate

Adherence to the Mediterranean diet (MEDAS-14)

Secondary outcomes:

Physical activity level (IPAQ-SF)

Tobacco and alcohol use

Self-esteem (Rosenberg Self-Esteem Scale)

Emotional intelligence (TMMS-24)

Health-related quality of life (SF-12, EQ-VAS)

Body image perception and risk of disordered eating (SCOFF)

Ethical Considerations

The study was approved by the Galician Clinical Research Ethics Committee (Ref. 2016/567), and all participants provided written informed consent.

ELIGIBILITY:
Inclusion Criteria:

Adults aged between 18 and 65 years.

Members of the university community (students, academic staff, or administrative personnel) enrolled in the University Sports Service.

Willingness to participate in the 4-month supervised physical activity and health education program.

Ability to provide written informed consent.

Exclusion Criteria:

Presence of any medical condition that contraindicates physical exercise (e.g., unstable cardiovascular disease, severe musculoskeletal injury, or uncontrolled hypertension).

Current participation in another structured exercise or nutrition program.

Pregnancy.

Inability to attend at least 75% of scheduled sessions.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 159 (Actual)
Dates: Start 2016-09-01 (Actual); Primary Completion 2017-06-30 (Actual); Study Completion 2017-07-31 (Actual)

PRIMARY OUTCOMES:
Change in Systolic and Diastolic Blood Pressure (SBP and DBP) | Baseline and Month 4
  Mean change in systolic and diastolic blood pressure (mmHg) from baseline to 4 months.
Change in Body Mass Index (BMI) | Baseline and Month 4
  Mean change in participants' body mass index (BMI, kg/m²) from baseline to 4 months, comparing the supervised intervention group and the control group.
Change in Resting Heart Rate (HR) | Baseline and Month 4
  Mean change in resting heart rate (beats per minute) from baseline to 4 months.
Change in Adherence to the Mediterranean Diet (MEDAS-14 score) | Baseline and Month 4
  Change in adherence to the Mediterranean diet assessed using the 14-item MEDAS questionnaire.

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared because the dataset contains personal health and academic information collected under institutional confidentiality agreements. De-identified summary data supporting the findings are available from the corresponding author upon reasonable request.

REFERENCES:
- [Background] Ware J Jr, Kosinski M, Keller SD. A 12-Item Short-Form Health Survey: construction of scales and preliminary tests of reliability and validity. Med Care. 1996 Mar;34(3):220-33. doi: 10.1097/00005650-199603000-00003. PMID 8628042
- [Background] Craig CL, Marshall AL, Sjostrom M, Bauman AE, Booth ML, Ainsworth BE, Pratt M, Ekelund U, Yngve A, Sallis JF, Oja P. International physical activity questionnaire: 12-country reliability and validity. Med Sci Sports Exerc. 2003 Aug;35(8):1381-95. doi: 10.1249/01.MSS.0000078924.61453.FB. PMID 12900694
- [Background] Salovey P, Mayer JD, Goldman SL, Turvey C, Palfai TP. Emotional attention, clarity, and repair: exploring emotional intelligence using the Trait Meta-Mood Scale. In: Pennebaker JW, editor. Emotion, disclosure, and health. Washington, DC: American Psychological Association; 1995. p. 125-54.
- [Background] Schroder H, Fito M, Estruch R, Martinez-Gonzalez MA, Corella D, Salas-Salvado J, Lamuela-Raventos R, Ros E, Salaverria I, Fiol M, Lapetra J, Vinyoles E, Gomez-Gracia E, Lahoz C, Serra-Majem L, Pinto X, Ruiz-Gutierrez V, Covas MI. A short screener is valid for assessing Mediterranean diet adherence among older Spanish men and women. J Nutr. 2011 Jun;141(6):1140-5. doi: 10.3945/jn.110.135566. Epub 2011 Apr 20. PMID 21508208
- [Background] Sánchez A, et al. Adherence to the Mediterranean diet in a university population: factors associated and relationship with body composition. Nutr Hosp. 2017;34(5):1174-81.
- [Background] Práxedes A, et al. Nivel de actividad física y factores de riesgo cardiovascular en universitarios. Retos. 2016;30:157-61.